CLINICAL TRIAL: NCT03387163
Title: PROVIDE-HF: Patient Reported Outcomes inVestigation Following Initiation of Drug Therapy With Entresto (Sacubitril/Valsartan) in Heart Failure
Brief Title: Patient Reported Outcomes inVestigation Following Initiation of Drug Therapy With Entresto (Sacubitril/Valsartan) in Heart Failure
Acronym: PROVIDE-HF
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BUS17
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure, Systolic
Keywords: Heart failure; Reduced left ventricular ejection fraction; Chronic Systolic Heart failure; Sacubitril /Valsartan; Patient reported outcomes (PRO); Kansas City Cardiomyopathy Questionnaire (KCCQ); Patient Centered Outcomes Research Network (PCORNeT); Common Data Model (CDM)
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sacubitril/Valsartan: Chronic systolic heart failure patients newly prescribed in mg. twice daily.
  Interventions: Drug: Sacubitril/Valsartan
- ACEi/ARB: Chronic systolic heart failure patients receiving ACEi/ARB and no s/v

INTERVENTIONS:
Drug: Sacubitril/Valsartan — commercially available Sacubitril/Valsartan: 24/26; 49/51 ; 97/103
  Groups: Sacubitril/Valsartan

SUMMARY:
Real-world evidence of the clinical course of patient symptoms following initiation of sacubitril/valsartan via PROs with a patient-centered study design will provide important evidence of potentially beneficial outcomes associated with the use of this therapy.

DETAILED DESCRIPTION:
This is a prospective cohort study of 400 chronic HF patients that will also examine and describe retrospective electronic health record data. We will use the PCORnet (Patient Centered Outcomes Research Network, see "data sources" below) infrastructure to (1) identify a cohort of chronic systolic HF patients initiated on sacubitril/valsartan (N=200) as well as a comparator group of similar HF patients not initiated on sacubitril/valsartan (N=200) but with background ACE/ARB therapy and (2) evaluate baseline and follow-up PROs via an electronic patient reported outcomes (ePRO) form in the eCOS database for 12 weeks.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of chronic systolic HF
* Active care by a provider in a healthcare system connected to a PCORnet data partner
* Ability to speak and read English (given the use of the English ePRO technology)
* Newly initiating sacubitril/valsartan (observational sacubitril/valsartan treatment group only - within 1 week of first dose)
* At least a 25% change ACE/ARB dose (including increase and decrease; or initiation or medication switching to another ACEI/ARB) in the last 6 months (comparator group only)
* Reliable access to the internet

Exclusion criteria:

* Inability to provide informed consent
* Life expectancy < 6 months
* For comparator group patients: Physician documentation of planned initiation of sacubitril/valsartan within 12 weeks

Other protocol inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 adult patients with chronic systolic HF in PCORnet. We will focus on chronic systolic HF patients initiated on sacubitril/valsartan and a comparator group not initiated on sacubitril/valsartan sacubitril (but with background ACE/ARB therapy and recent titration of these medications).
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 12 weeks in the KCCQ | Baseline to weeks 2, 4, 8 and 12
  Kansas City Cardiomyopathy Questionnaire (KCCQ) - self-administered, 23-item questionnaire that quantifies physical limitations, symptoms, self-efficacy, social interference and quality of life in patients with heart failure.

SECONDARY OUTCOMES:
Responder analysis for a 5-point improvement in KCCQ to week 12 | Baseline to week 12
  Binary response for a 5-point improvement in KCCQ to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mentz RJ, Xu H, O'Brien EC, Thomas L, Alexy T, Gupta B, Vilaro J, Lala A, DeVore AD, Dhingra R, Briasoulis A, Simon MA, Stehlik J, Rodgers JE, Dunlay SM, Abshire M, Wells QS, Barringhaus KG, Eckman PM, Lowes BD, Espinoza J, Blanco R, Shen X, Duffy CI, Hernandez AF. PROVIDE-HF primary results: Patient-Reported Outcomes inVestigation following Initiation of Drug therapy with Entresto (sacubitril/valsartan) in heart failure. Am Heart J. 2020 Dec;230:35-43. doi: 10.1016/j.ahj.2020.09.012. Epub 2020 Sep 24. PMID 32980364